CLINICAL TRIAL: NCT02004873
Title: Micra Transcatheter Pacing Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Micra
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Results first posted 2017-01-05 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2017-12

CONDITIONS: Class I or II Indication for Implantation of a Single Chamber Ventricular Pacemaker According to ACC/AHA/HRS 2001 Guidelines and Any National Guidelines
Keywords: pacemaker; leadless; single chamber

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Micra Pacemaker Implant (Experimental)
  Interventions: Device: Micra Pacemaker Implant

INTERVENTIONS:
Device: Micra Pacemaker Implant

SUMMARY:
The purpose of this clinical study is to evaluate the safety and efficacy of the Micra Transcatheter Pacing System and to assess long term performance.

DETAILED DESCRIPTION:
The study is being conducted in 56 sites located around the world, including 30 sites in the United States (U.S.).

Up to 780 subjects were planned to be enrolled (i.e. consented) to allow up to 720 subjects to be implanted enabling at least 600 subjects to be followed for at least 12-months post-implant.

There are two primary objectives in this study (one safety and one efficacy). The primary safety objective of the study is to evaluate major complications related to the Micra system or procedure. The primary safety endpoint was pre-specified to be evaluated at 6-months (183 days) post-implant. The primary efficacy objective, Micra pacing capture thresholds, was also pre-specified to be evaluated six months post-implant. This study also has a separate long term safety objective that will provide additional long-term safety data following potential regulatory submissions.

All subjects will be followed until official study closure (official study closure is defined as when Medtronic and/or FDA requirements have been satisfied per the Clinical Investigational Plan and/or by a decision by Medtronic or regulatory authority).

Additionally, the Micra Accelerometer Sensor Sub-Study (MASS) is being conducted at 4 centers already active in the Micra study in Austria, Spain, Hungary and France. Forty (40) subjects were enrolled in the Sub-Study, and enrollment in the Sub-Study was complete as of March 31, 2016. The purpose of the Sub-Study is to test feasibility for future enhancements in the Micra device functionalities.

An algorithm was designed to sense the atrial contraction using the Micra accelerometer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have a Class I or II indication for implantation of a single chamber ventricular pacemaker according to ACC/AHA/HRS 2008 guidelines and any national guidelines
* Subjects who are able and willing to undergo the study requirements and are expected to be geographically stable for the duration of the follow-up.
* Subjects who are at least 18 years of age (or older, if required by local law).

Exclusion Criteria:

* Subjects who are entirely pacemaker dependent (escape rhythm <30 bpm). (Please note: Subjects who are entirely pacemaker dependent (escape rhythm <30 bpm) can now be included in the study. Medtronic notified all sites on July 23, 2014 that the restriction against pacemaker dependent subjects was lifted, following review of the Early Performance Assessment.)
* Subject has an existing or prior pacemaker, ICD or CRT device implant.
* Subject has unstable angina pectoris or has had an acute myocardial infarction (AMI) in the 30 days prior to eligibility assessment.
* Subjects with current implantation of neurostimulator or any other chronically implanted device which uses current in the body. Note that a temporary pacing wire is allowed.
* Subjects with a mechanical tricuspid valve, implanted vena cava filter, or left ventricular assist device (LVAD).
* Subjects who are morbidly obese and physician believes telemetry communication of ≤5 inches (12.7 cm) could not be obtained with programmer head.
* Subjects whose femoral venous anatomy is unable to accommodate a 23 French introducer sheath or implant on the right side of the heart (for example, due to obstructions or severe tortuosity) in the opinion of the implanter.
* Subjects who are considered as unable to tolerate an urgent sternotomy
* Subjects with a known intolerance to Nickel-Titanium (Nitinol) Alloy.
* Subjects for whom a single dose of 1.0mg dexamethasone acetate may be contraindicated.
* Subjects with a life expectancy of less than 12- months.
* Subjects who are currently enrolled or planning to participate in a potentially confounding drug or device trial during the course of this study. Coenrollment in concurrent trials is only allowed when document pre-approval is obtained from the Medtronic study manager.
* Pregnant women, or women of child bearing potential and who are not on a reliable form of birth control.
* Subjects with exclusion criteria required by local law (e.g. age, breast feeding, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 744 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dwight Reynolds, Study Chair — University of Oklahoma; Philippe Ritter, Study Chair — Hôpital Haut-Lévêque
Locations (56):
- United States (30):
  - Scripps, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Baptist Heart Specialists, Jacksonville, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Iowa Heart Center, West Des Moines, Iowa
  - Michigan Heart, Ypsilanti, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - CentraCare Heart & Vascular Center, Saint Cloud, Minnesota
  - Mid America Heart Institute, Kansas City, Missouri
  - Morristown Memorial Hospital, Morristown, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - North Shore LIJ Health System, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - University of Oklahoma Health Science Center (OUHSC), Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Providence Health & Services, Portland, Oregon
  - Lancaster Heart & Vascular Research Institute, Lancaster, Pennsylvania
  - University of Pittsburgh Medical Center UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - The Stern Cardiovascular Clinic, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Research Institute, Dallas, Texas
  - St. Luke's Medical Center, Houston, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Aurora Cardiovascular Services, Milwaukee, Wisconsin
- Princess Alexandria Hospital, Woolloongabba, Queensland, Australia
- Allgemeines Krankenhaus der Stadt Linz, Linz, Austria
- Canada (2):
  - Montreal Heart Institute, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec (IUCPQ), Québec
- Fuwai Hospital Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China
- Nemocnice Na Homolce, Prague, Czechia
- Rigshospitalet, Copenhagen, Denmark
- Hôpital Haut-Lévêque - CHU de Bordeaux, Bordeaux, France
- University General Hospital of Heraklion, Heraklion, Greece
- Magyar Honvédség Honvédkorház, Budapest, Hungary
- India (3):
  - CARE Hospitals, Hyderabad
  - All India Institute of Medical Sciences, New Delhi
  - Govind Ballabh Pant Hospital, New Delhi
- Azienda Ospedaliero Universitaria Pisana - Stabilimento Santa Chiara, Pisa, Italy
- Japan (4):
  - National Cerebral and Cardiovascular Center, Osaka
  - Showa University Hospital, Shinagawa-Ku
  - Kyorin University Hospital, Tokyo
  - Yokohama City University Hospital, Yokohama
- Institut Jantung Negara - National Heart Institute, Kuala Lumpur, Malaysia
- Netherlands (3):
  - Academisch Medisch Centrum (AMC), Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - St. Antonius Ziekenhuis - Locatie Nieuwegein, Nieuwegein
- Klinicki Centar Srbije, Belgrade, Serbia
- Groote Schuur Hospital, Cape Town, South Africa
- Hospital Universitari Clínic de Barcelona, Barcelona, Spain
- Southampton General Hospital - University Hospital Southampton NHS Foundation Trust, Southampton, United Kingdom

REFERENCES:
- [Derived] Piccini JP, Cunnane R, Steffel J, El-Chami MF, Reynolds D, Roberts PR, Soejima K, Steinwender C, Garweg C, Chinitz L, Ellis CR, Stromberg K, Fagan DH, Mont L. Development and validation of a risk score for predicting pericardial effusion in patients undergoing leadless pacemaker implantation: experience with the Micra transcatheter pacemaker. Europace. 2022 Jul 21;24(7):1119-1126. doi: 10.1093/europace/euab315. PMID 35025987
- [Derived] El-Chami MF, Shinn T, Bansal S, Martinez-Sande JL, Clementy N, Augostini R, Ravindran B, Sagi V, Ramanna H, Garweg C, Roberts PR, Soejima K, Stromberg K, Fagan DH, Zuniga N, Piccini JP. Leadless pacemaker implant with concomitant atrioventricular node ablation: Experience with the Micra transcatheter pacemaker. J Cardiovasc Electrophysiol. 2021 Mar;32(3):832-841. doi: 10.1111/jce.14881. Epub 2021 Jan 23. PMID 33428248
- [Derived] Garg A, Koneru JN, Fagan DH, Stromberg K, Padala SK, El-Chami MF, Roberts PR, Piccini JP, Cheng A, Ellenbogen KA. Morbidity and mortality in patients precluded for transvenous pacemaker implantation: Experience with a leadless pacemaker. Heart Rhythm. 2020 Dec;17(12):2056-2063. doi: 10.1016/j.hrthm.2020.07.035. Epub 2020 Aug 4. PMID 32763431
- [Derived] Tjong FVY, Beurskens NEG, de Groot JR, Waweru C, Liu S, Ritter P, Reynolds D, Wilde AAM, Knops RE; Micra Investigators. Health-related quality of life impact of a transcatheter pacing system. J Cardiovasc Electrophysiol. 2018 Dec;29(12):1697-1704. doi: 10.1111/jce.13726. Epub 2018 Oct 15. PMID 30168233
- [Derived] El-Chami MF, Al-Samadi F, Clementy N, Garweg C, Martinez-Sande JL, Piccini JP, Iacopino S, Lloyd M, Vinolas Prat X, Jacobsen MD, Ritter P, Johansen JB, Tondo C, Liu F, Fagan DH, Eakley AK, Roberts PR. Updated performance of the Micra transcatheter pacemaker in the real-world setting: A comparison to the investigational study and a transvenous historical control. Heart Rhythm. 2018 Dec;15(12):1800-1807. doi: 10.1016/j.hrthm.2018.08.005. Epub 2018 Aug 10. PMID 30103071
- [Derived] Okabe T, El-Chami MF, Lloyd MS, Buck B, Gornick CC, Moore JC, Augostini RS, Hummel JD. Leadless pacemaker implantation and concurrent atrioventricular junction ablation in patients with atrial fibrillation. Pacing Clin Electrophysiol. 2018 May;41(5):504-510. doi: 10.1111/pace.13312. Epub 2018 Apr 16. PMID 29476660
- [Derived] Soejima K, Asano T, Ishikawa T, Kusano K, Sato T, Okamura H, Matsumoto K, Taguchi W, Stromberg K, Lande J, Kobayashi Y; Micra Transcatheter Pacing Study Group. Performance of Leadless Pacemaker in Japanese Patients vs. Rest of the World - Results From a Global Clinical Trial. Circ J. 2017 Oct 25;81(11):1589-1595. doi: 10.1253/circj.CJ-17-0259. Epub 2017 May 30. PMID 28566657
- [Derived] Lloyd M, Reynolds D, Sheldon T, Stromberg K, Hudnall JH, Demmer WM, Omar R, Ritter P, Hummel J, Mont L, Steinwender C, Duray GZ. Rate adaptive pacing in an intracardiac pacemaker. Heart Rhythm. 2017 Feb;14(2):200-205. doi: 10.1016/j.hrthm.2016.11.016. Epub 2016 Nov 15. PMID 27871854
- [Derived] Reynolds D, Duray GZ, Omar R, Soejima K, Neuzil P, Zhang S, Narasimhan C, Steinwender C, Brugada J, Lloyd M, Roberts PR, Sagi V, Hummel J, Bongiorni MG, Knops RE, Ellis CR, Gornick CC, Bernabei MA, Laager V, Stromberg K, Williams ER, Hudnall JH, Ritter P; Micra Transcatheter Pacing Study Group. A Leadless Intracardiac Transcatheter Pacing System. N Engl J Med. 2016 Feb 11;374(6):533-41. doi: 10.1056/NEJMoa1511643. Epub 2015 Nov 9. PMID 26551877
- [Derived] Ritter P, Duray GZ, Steinwender C, Soejima K, Omar R, Mont L, Boersma LV, Knops RE, Chinitz L, Zhang S, Narasimhan C, Hummel J, Lloyd M, Simmers TA, Voigt A, Laager V, Stromberg K, Bonner MD, Sheldon TJ, Reynolds D; Micra Transcatheter Pacing Study Group. Early performance of a miniaturized leadless cardiac pacemaker: the Micra Transcatheter Pacing Study. Eur Heart J. 2015 Oct 1;36(37):2510-9. doi: 10.1093/eurheartj/ehv214. Epub 2015 Jun 4. PMID 26045305
- [Derived] Ritter P, Duray GZ, Zhang S, Narasimhan C, Soejima K, Omar R, Laager V, Stromberg K, Williams E, Reynolds D; Micra Transcatheter Pacing Study Group. The rationale and design of the Micra Transcatheter Pacing Study: safety and efficacy of a novel miniaturized pacemaker. Europace. 2015 May;17(5):807-13. doi: 10.1093/europace/euv026. Epub 2015 Apr 7. PMID 25855677

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled 744 subjects at 56 centers in 19 countries worldwide between December 2013 and May 2015.
Pre-assignment Details: Of the 744 subjects enrolled, 19 exited from the study without attempting Micra implant (7 did not meet inclusion / exclusion criteria, 12 due to other miscellaneous reasons), 6 attempted Micra implant but were unsuccessful, and the remaining 719 subjects were successfully implanted with a Micra device.
Groups:
- Micra Pacemaker Implant: All subjects who attempted Micra implant procedure
Period: Overall Study
Arm/Group | Micra Pacemaker Implant
Started | 725 (Micra Implant Attempt)
Micra Implant Success | 719
Completed | 301 (6-Month Follow-up)
Not Completed | 424
Not completed — Implant unsuccessful | 6
Not completed — Awaiting 6-month visit | 390
Not completed — Missed 6-month visit | 4
Not completed — Death | 23
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All subjects enrolled in the study
Groups:
- Micra Study Enrollments: All subjects enrolled in the Micra study
Arm/Group | Micra Study Enrollments
Number analyzed (Participants) | 744
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.7 (11.0)
Sex/Gender, Customized [Number; unit: participants]
  Female | 309
  Male | 434
  Missing | 1
Region of Enrollment [Number; unit: participants]
  Hungary | 56
  United States | 297
  Japan | 38
  United Kingdom | 30
  Malaysia | 21
  Spain | 54
  India | 19
  Greece | 5
  Canada | 15
  Austria | 50
  Czech Republic | 43
  Netherlands | 37
  China | 7
  Denmark | 3
  Italy | 17
  South Africa | 3
  Serbia | 7
  France | 38
  Australia | 4

OUTCOME MEASURES:

1. Primary Outcome: Major Complications
Description: Micra system and/or procedure related major complication free rate at 6-months post-implant.
Time Frame: Implant to 6 Months Post Implant
Population: All subjects who attempted Micra implant procedure
Measure: Number (98.66% Confidence Interval); unit: Kaplan-Meier survival probability (%)
Arm/Group | Micra Pacemaker Implant
Number analyzed (Participants) | 725
Kaplan-Meier survival probability (%) | 96.0 [93.3 to 97.6]
Statistical Analysis 1: Comparison: Micra Pacemaker Implant; Null hypothesis: Major complication free rate at 6 months post-implant is less than or equal to 83%. Alternative hypothesis: Major complication free rate at 6 months post-implant is greater than 83%; Test type: Superiority or Other; p < 0.0001, z-test, 1-sided — The threshold for statistical significance was 0.0067, determined by the pre-specified alpha spending function for the interim analysis; Kaplan-Meier survival probability (%) = 96.0, 98.66% CI 2-sided [93.3 to 97.6] — The major complication free rate (i.e. survival probability) was estimated using the Kaplan-Meier method. The coverage level for the confidence interval was 98.66%, determined by the pre-specified alpha spending function for the interim analysis

2. Primary Outcome: Pacing Capture Threshold
Description: Subjects that have an adequate pacing capture threshold (PCT) at the 6-month post-implant visit, which is defined as PCT <=2 volts at 0.24 ms pulse width and the increase in PCT from implant to 6 months <=1.5 volts. The pacing capture threshold is the minimal electrical stimulus required to produce consistent cardiac depolarization. It is the minimum amount of energy that is required for a pacemaker to pace the heart.
Time Frame: 6 Months Post Implant
Population: Subjects implanted with Micra who had paired implant and 6-month auto decrement PCT values (at 0.24 ms), or who had a system modification or alternative device implant prior to 6 months due to elevated threshold.
Measure: Number; unit: participants
Groups:
- Micra Subjects With Implant and 6-month PCT Data: Subjects implanted with Micra who had paired implant and 6-month auto decrement PCT values (0.24 ms), or who had a system modification or alternative device implant prior to 6 months due to elevated threshold.
Arm/Group | Micra Subjects With Implant and 6-month PCT Data
Number analyzed (Participants) | 297
participants | 292
Statistical Analysis 1: Comparison: Micra Subjects With Implant and 6-month PCT Data; Null hypothesis: Percentage of subjects with an adequate pacing capture threshold at 6-months post-implant is less than or equal to 80%. Alternative hypothesis: Percentage of subjects with an adequate pacing capture threshold at 6-months post-implant is greater than 80%; Test type: Superiority or Other; p < 0.0001, Exact Binomial test — [p-value comment as in outcome 1, analysis 1]; Percentage of subjects (%) = 98.3, 98.66% CI 2-sided [95.4 to 99.6] — The coverage level for confidence interval was 98.66%, determined by the pre-specified alpha spending function for the interim analysis

3. Secondary Outcome: Ventricular Capture Management Threshold
Description: Subjects that have a ventricular capture management threshold (VCMT) that is within 0.5 Volts of the manual (auto decrement) PCT (at 0.24 ms pulse width) at the 6-month post-implant visit. The VCMT is an automatically measured pacing capture threshold that is measured by the Micra device's pacing algorithm. In contrast, the manual (auto decrement) pacing capture threshold is measured by the clinician during a study visit.
Time Frame: 6 Months Post Implant
Population: Subjects implanted with Micra who had paired ventricular capture management PCT and auto decrement PCT data available at the 6-month visit.
Measure: Number; unit: participants
Groups:
- Micra Subjects With 6-month PCT Data: Subjects implanted with Micra who had paired ventricular capture management PCT and auto decrement PCT data available at the 6-month visit.
Arm/Group | Micra Subjects With 6-month PCT Data
Number analyzed (Participants) | 280
participants | 279
Statistical Analysis 1: Comparison: Micra Subjects With 6-month PCT Data; Null hypothesis: Percentage of subjects with VCMT within 0.5 Volts of auto decrement PCT at 6 months post-implant is less than or equal to 85%. Alternative hypothesis: Percentage of subjects with VCMT within 0.5 Volts of auto decrement PCT at 6 months post-implant is greater than 85%; Test type: Superiority or Other; p < 0.0001, Exact Binomial test — Holm adjustment for multiple comparisons for secondary objectives was used. The threshold for statistical significance was 0.0067, determined by the pre-specified alpha spending function for the interim analysis; Percentage of subjects (%) = 99.6, 98.66% CI 2-sided [97.5 to 100.0] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Rate Response Operation of Micra
Description: Assessment of whether the Micra sensor-indicated rate derived from the input of the accelerometer during the Minnesota Pacemaker Response Exercise Protocol (M-PREP) treadmill test conducted at the 3-month and 6-month follow-up visits was proportional to the workload. The sensor-indicated rate (in min^-1) and workload (in METS) were normalized for each subject relative to their minimum and maximum possible values so the normalized values have a minimum possible value of zero and a maximum possible value of 1. These normalized values were used in a random effect linear regression model to assess the relationship between the sensor-indicated rate and workload via estimation of the Kay-Wilkoff slope parameter. The tests at 3-month and 6-month visits were combined in one analysis.
Time Frame: 3 Months and 6 Months Post Implant (combined analysis)
Population: Subjects implanted with Micra who had usable M-PREP test(s) at 3-month and/or 6-month visits.
Measure: Mean (90% Confidence Interval); unit: regression slope parameter
Units Other Than Participants: M-PREP tests
Groups:
- Micra Subjects With Usable M-PREP Data: Subjects implanted with Micra who had usable M-PREP test(s) at 3-month and/or 6-month visits.
Arm/Group | Micra Subjects With Usable M-PREP Data
Number analyzed (Participants) | 20
Number analyzed (M-PREP tests) | 30
regression slope parameter | 0.864 [0.768 to 0.961]
Statistical Analysis 1: Comparison: Micra Subjects With Usable M-PREP Data; Null hypothesis: Kay-Wilkoff slope parameter is < 0.65 or > 1.35 Alternative hypothesis: Kay-Wilkoff slope parameter is between 0.65 and 1.35; Test type: Non-Inferiority or Equivalence — The equivalence margin is 0.35. The Micra sensor indicated rate is considered proportional to the workload if the 90% CI for the Kay-Wilkoff slope parameter falls into [0.65, 1.35]; p < 0.001, t-test, 1 sided — Holm adjustment for multiple comparisons for secondary objectives was used. Two One-sided Test (TOST) procedure was used at the 0.05 significance level; Two One-sided Test (TOST); Slope = 0.864, 90% CI 2-sided [0.768 to 0.961] — A random effect linear regression model was used to assess if the Micra sensor-indicated rate was proportional to the workload using the Kay-Wilkoff model. The Kay-Wilkoff slope parameter was estimated along with its 90% CI

ADVERSE EVENTS:
Time Frame: From implant attempt to last subject follow-up, ranging from 0 to 14.5 months
Arm/Group | Micra Pacemaker Implant
Serious Adverse Events (participants affected / at risk) | 226/725
Other Adverse Events (participants affected / at risk) | 0/725
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Micra Pacemaker Implant (N=725)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 6 (6)
Angina pectoris (Cardiac disorders) | 4 (4)
Angina unstable (Cardiac disorders) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 13 (13)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 5 (5)
Bundle branch block right (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 52 (64)
Cardiac perforation (Cardiac disorders) | 3 (3)
Coronary artery disease (Cardiac disorders) | 5 (5)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 11 (11)
Pericarditis (Cardiac disorders) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Tachycardia induced cardiomyopathy (Cardiac disorders) | 1 (1)
Torsade de pointes (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 3 (3)
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Coronary artery restenosis (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Device dislocation (General disorders) | 1 (1)
Device pacing issue (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 8 (8)
Pacemaker syndrome (General disorders) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Arthritis bacterial (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2)
Bronchopneumonia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3)
Clostridium difficile infection (Infections and infestations) | 2 (2)
Endocarditis (Infections and infestations) | 2 (2)
Epiglottitis (Infections and infestations) | 1 (1)
Gastritis viral (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Infected seroma (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 3 (3)
Neutropenic sepsis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 19 (19)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 6 (6)
Septic shock (Infections and infestations) | 3 (4)
Sinusitis (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 8 (8)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1)
Cardiac valve rupture (Injury, poisoning and procedural complications) | 1 (1)
Dialysis related complication (Injury, poisoning and procedural complications) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 3 (3)
Laceration (Injury, poisoning and procedural complications) | 2 (2)
Medication error (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
International normalised ratio increased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Axillary mass (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Cognitive disorder (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2)
Dementia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 8 (8)
Syncope (Nervous system disorders) | 7 (7)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 4 (4)
Renal failure chronic (Renal and urinary disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 3 (3)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Incisional drainage (Surgical and medical procedures) | 2 (2)
Accelerated hypertension (Vascular disorders) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 5 (5)
Circulatory collapse (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3)
Embolism (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (4)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 6 (6)
Ischaemia (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Temporal arteritis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, contracts allow investigators to publish study results per the protocol and publication plan. Investigators and Participating Institutions will provide any publication of Study Data generated by PI and/or Participating Institution to Medtronic for review prior to submission to determine if confidential information ("CI") is included and to check for technical correctness. Medtronic may not censor/interfere with the publication beyond the extent necessary to protect CI.